CLINICAL TRIAL: NCT02048670
Title: A Pilot Project to Investigate the Use of an External Vestibular Prosthesis Potential to Improve Clinical Management of Chronic Subjective Dizziness (CSD)
Brief Title: Pilot Project on External Vestibular Prosthesis in Chronic Subjective Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey P. Staab, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-005525
Record Dates: First submitted 2014-01-22; First posted 2014-01-29 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Dizziness Chronic
Keywords: Pilot study; Assessment of sway phase; Therapy trial phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Subjective Dizziness Syndrome Subjects (Experimental): Subjects diagnosed with Chronic Subjective Dizziness Syndrome (CDS) will wear the BalanceBelt while performing test involving walking and balance.
  Interventions: Device: Balance Belt
- Healthy Subjects (Active Comparator): Age matched healthy subjects without complaints of balance or dizziness problems will wear the BalanceBelt while performing test involving walking and balance.
  Interventions: Device: Balance Belt

INTERVENTIONS:
Device: Balance Belt — Vestibular habituation therapy worn under the clothes around the waist that uses sensitive motion detectors and vibrates against the skin at four locations to provide information about posture and gait
  Other Names: Stabalon Belt; Vibrating Belt

SUMMARY:
Researchers are gathering information on the safety and effectiveness of a new device called the BalanceBelt.

DETAILED DESCRIPTION:
Ten consecutive subjects, ages 25-70 years, diagnosed with Chronic Subjective Dizziness (CDS) and ten healthy age and gender matched subjects will be asked to perform tests involving walking and balance while wearing the BalanceBelt. The BalanceBelt is a lightweight belt that will be worn under the clothes around the subjects waist and uses sensitive motion detectors and vibrates against the skin at four locations to provide information about posture and motion.

ELIGIBILITY:
Subject population: 20 patients with diagnosis of Chronic Subjective Dizziness (CSD) and 10 normal volunteers.

Inclusion Criteria:

* Subjects will be 25-70 years of age inclusive and pregnant women may participate.
* Patients will have CSD as their primary diagnosis for the cause of their balance and dizziness complaints provided by the Behavioral Medicine Program for Dizziness, a division of the Department of Psychiatry & Psychology.
* Normal volunteers will have a negative history of otologic & neurologic disorders and no history of dizziness and balance problems.
* Normal volunteers will have normal findings on a screening office examination for peripheral and central vestibular system involvement (see methods for details of the examination) and screening for normal or symmetrical hearing loss of explainable origin.

Exclusion Criteria:

* Patients with positive indications from testing of peripheral and/or central vestibular system involvement that is felt to be influencing the symptoms reported beyond the CSD alone.
* Patients with mobility restriction that would prevent participating in the tests or the intensive therapy trials.
* Subjects with hearing impairment that interferes with oral communication.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Staab, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Subjective Dizziness Syndrome Subjects | Healthy Subjects
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Subjective Dizziness Syndrome Subjects | Healthy Subjects | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.2) | 56.3 (11.6) | 56.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Degrees of Sway
Description: The Sensory Organization Test is a six condition standard evaluation of balance control performed on a dynamic platform that can record sway movement in the A/P dimension while the sensory inputs from proprioception and vision are varied though the platform and visual surround movements. Condition 1 - eyes open, visual locked, platform locked. Condition 2 - eyes closed, visual locked, platform locked. Condition 3 - eyes open, visual unlocked, platform locked. Condition 4 - eyes open, visual locked, platform unlocked. Condition 5 - eyes closed, visual locked, platform unlocked. Condition 6 - eyes open, visual unlocked, platform unlocked. All participants progress though the exam, starting with condition 1 and ending with condition 6. All conditions were completed two to three times depending on performance with the average of each condition reported.
Time Frame: baseline
Measure: Mean (Standard Error); unit: degrees of sway
Arm/Group | Chronic Subjective Dizziness Syndrome Subjects | Healthy Subjects
Number analyzed (Participants) | 6 | 6
degrees of sway
  Condition 1 | 1.824 (0.266) | 0.746 (0.278)
  Condition 2 | 1.638 (0.259) | 0.573 (0.287)
  Condition 3 | 1.605 (0.252) | 0.869 (0.278)
  Condition 4 | 1.480 (0.259) | 1.979 (0.259)
  Condition 5 | 1.900 (0.270) | 1.892 (0.278)
  Condition 6 | 1.519 (0.274) | 2.666 (0.274)
Statistical Analysis 1: Comparison: Chronic Subjective Dizziness Syndrome Subjects vs Healthy Subjects; Condition 1 - eyes open, visual surround locked, platform locked; Test type: Superiority; p = 0.005, Kruskal-Wallis
Statistical Analysis 2: Comparison: Chronic Subjective Dizziness Syndrome Subjects vs Healthy Subjects; Condition 2 - eyes closed, visual surround locked, platform locked; Test type: Superiority; p = 0.006, Kruskal-Wallis
Statistical Analysis 3: Comparison: Chronic Subjective Dizziness Syndrome Subjects vs Healthy Subjects; Condition 3 - eyes open, visual surround unlocked, platform locked; Test type: Superiority; p = 0.051, Kruskal-Wallis
Statistical Analysis 4: Comparison: Chronic Subjective Dizziness Syndrome Subjects vs Healthy Subjects; Condition 4 - eyes open, visual surround locked, platform unlocked; Test type: Superiority; p = 0.173, Kruskal-Wallis
Statistical Analysis 5: Comparison: Chronic Subjective Dizziness Syndrome Subjects vs Healthy Subjects; Condition 5 - eyes closed, visual surround locked, platform unlocked; Test type: Superiority; p = 0.985, Kruskal-Wallis
Statistical Analysis 6: Comparison: Chronic Subjective Dizziness Syndrome Subjects vs Healthy Subjects; Condition 6 - eyes open, visual surround unlocked, platform unlocked; Test type: Superiority; p = 0.003, Kruskal-Wallis

2. Secondary Outcome: Visual Analog Scales Score
Description: For the therapy portion of the study aim #2 Visual Analog Scales (VAS) related to the intensity of symptoms provoked by visual motion, head movements and walking in visually complex environments. The average Visual Analog Scale scores for the patient group pre and post therapy will be compared for any significant difference in the score (p<0.05). The VAS ranges from 0-10, where 0 is no symptoms and 10 is the most intense symptoms experienced.
Time Frame: baseline
Population: This outcome measure was not evaluated in this study. No data have been collected for this outcome measure.
Arm/Group | Chronic Subjective Dizziness Syndrome Subjects | Healthy Subjects
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: For this study, adverse events will be captured and reported from enrollment to the end of the study treatment for each subject, approximately one day.
Arm/Group | Chronic Subjective Dizziness Syndrome Subjects | Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT02048670/Prot_SAP_000.pdf